CLINICAL TRIAL: NCT05105321
Title: Efficacy and Safety of Berberine on Primary Prevention of Cardiovascular Diseases and Diabetes in Metabolic Syndrome: a Randomized, Controlled Trial
Brief Title: Cardiovascular Diseases and Diabetes Prevention Programme in Metabolic Syndrome (CDPP)
Acronym: CDPP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tang Yida (Other)
Collaborators: Chinese Society of Cardiology (Other)
Responsible Party: Sponsor-Investigator, Tang Yida, Chief-Cardiologist and Director, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CSCF2021A04
Record Dates: First submitted 2021-10-16; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Metabolic Syndrome
Keywords: Berberine; Cardiovascular Diseases; Diabetes; Metabolic Syndrome; Primary Prevention
MeSH Terms: conditions — Metabolic Syndrome; Cardiovascular Diseases; Diabetes Mellitus | interventions — Berberine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): Placebo plus healthy lifestyle intervention. Placebo with same appearance of berberine tablet will be orally taken twice daily and maintained until the last subject completes 3-year intervention.
  Interventions: Behavioral: Healthy lifestyle intervention
- Berberine Group (Experimental): Berberine plus healthy lifestyle intervention. Berberine dose is 500mg twice daily and maintained until the last subject completes 3-year intervention.
  Interventions: Drug: Berberine; Behavioral: Healthy lifestyle intervention

INTERVENTIONS:
Drug: Berberine — The tablet of berberine and placebo are both coated with white sugar and had the same appearance. Berberine tablet will be orally taken with a dose of 500mg twice daily
  Other Names: berberine hydrochloride
  Arms: Berberine Group
Behavioral: Healthy lifestyle intervention — Healthy lifestyle intervention will be launched according to the "Chinese guidelines on prevention of cardiovascular and metabolic diseases by Chinese Preventive Medical Association in 2019", including health lectures, health information promotion, health manual and so on.

SUMMARY:
The metabolic syndrome population is at high-risk of cardiovascular diseases and diabetes. How to effectively control the risk factors of this population is the key to primary prevention of cardiovascular diseases and diabetes in China. This study aims to explore the efficacy and safety of an intervention strategy with berberine that can effectively treat a variety of risk factors (hyperglycemia, dyslipidemia, hypertension).

DETAILED DESCRIPTION:
Metabolic syndrome (MS) is a condition with multiple abnormal metabolic components, including obesity, dysglycemia, dyslipidemia and hypertension. The components of metabolic syndrome are major risk factors for cardiovascular disease and diabetes. Cardiovascular disease (CVD) is the primary cause of death and disease burden in China. This study aims to explore an intervention drug that can effectively control a variety of risk factors (hyperglycemia, dyslipidemia, hypertension), so as to improve the effectiveness and practical feasibility of primary prevention. Berberine is a drug with multiple function. Basic studies and previous clinical studies suggest that it has definite regulatory effects on blood glucose, lipid levels and blood pressure with few adverse reactions. This study selected pleiotropic Berberine as a means of intervention. It would provide new thought and high-level evidence for the primary prevention of cardiovascular disease and diabetes in Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with metabolic syndrome aged 40-75 years old.
* Metabolic syndrome was defined according to the Chinese Guidelines for the Prevention and Treatment of Dyslipidemia in Adults (revised edition 2016). Subjects will be diagnosed with metabolic syndrome when meeting three or more of the following items: 1, central obesity and/or abdominal obesity (waist circumference ≥90cm for men and ≥ 85cm for women); 2, hyperglycemia (fasting blood glucose ≥6.10 mmol/L or two-hour blood glucose ≥7.80 mmol/L in glucose tolerance test); 3, hypertension: blood pressure ≥130/85 mmHg and/or diagnosed hypertension under treatment; 4, fasting triglyceride ≥1.7 mmol/L (150mg/dl); 5, fasting HDL cholesterol<1.0 mmol/L.

Exclusion Criteria:

* Previously diagnosed diabetes.
* Baseline LDL cholesterol≥130mg/dl (3.4mmol/L).
* Baseline triglyceride≥500mg/dl (5.6mmol/L).
* Baseline blood pressure ≥140/90 mmHg (twice not on the same day).
* Impaired liver function, have obvious clinical signs or symptoms of liver disease, acute or chronic hepatitis, alanine/aspartate aminotransferase levels >3 times the upper limit of the reference range at the screening visit.
* Renal dysfunction (glomerular filtration rate<45ml/min)
* Patients ventilated by ventilator.
* Hypersensitivity to berberine.
* Disease which may cause tissue hypoxia (especially acute disease, or worsening of chronic respiratory disease).
* Severe chronic gastrointestinal disease.
* Severe psychiatric illness.
* Cancer requiring treatment in past 5 years.
* Women who are pregnant or breastfeeding .
* Participation in another clinical trial within the past 30 days .
* Other significant disease that in the Investigator's opinion would exclude the subject from the trial.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5200 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Rate of composite cardiometabolic endpoints | three year
  The composite endpoints including cardiac death, nonfatal myocardial infarction, nonfatal stroke, and newly-diagnosed type 2 diabetes.

SECONDARY OUTCOMES:
Rate of composite endpoints of cardiovascular diseases 1 | three year
  The composite endpoints including cardiac death, nonfatal myocardial infarction, nonfatal stroke.
Rate of composite end point of cardiovascular disease 2 | three year
  The composite endpoints including cardiac death, nonfatal myocardial infarction, nonfatal stroke, successful resuscitation of cardiac arrest, heart failure, arterial revascularization.
Rates of each component of the composite end point | three year
  Each component of the composite end point
Rate of all-cause mortality | three year
  Death due to all causes.
Rate of newly diagnosed prediabetes | three year
  Prediabetes including impaired fasting glucose and abnormal glucose tolerance.
Rate of newly diagnosed hypertension | three year
  Hypertension is defined as blood pressure≥140/90 millimeters of mercury measured twice at not same day.
Rate of newly diagnosed malignancy | three year
  Newly diagnosed malignancy.
Concentrations of serum lipid parameters | three year
  Serum lipid parameters including total cholesterol, LDL cholesterol, HDL cholesterol, non-HDL cholesterol, triglycerides, Lp(a).
Changes of abdominal circumference | three year
  Measurement of abdominal circumference in centimeter
Changes of waist-hip ratio | three year
  Measurement of waist-hip ratio
Changes of body mass index | three year
  Measurement of body mass index in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Da Tang, MD, PhD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The data, analytic methods, and study materials will not be made available immediately to other researchers. The reason for the lack of availability is that we have signed an agreement with the sponsor to restrict approach to study data, and the access must be agreed by both investigator and sponsor. Request to get these materials can be sent to the corresponding author, and we will provide them to vetted and qualified applicants.

REFERENCES:
- [Background] Arnett DK, Blumenthal RS, Albert MA, Buroker AB, Goldberger ZD, Hahn EJ, Himmelfarb CD, Khera A, Lloyd-Jones D, McEvoy JW, Michos ED, Miedema MD, Munoz D, Smith SC Jr, Virani SS, Williams KA Sr, Yeboah J, Ziaeian B. 2019 ACC/AHA Guideline on the Primary Prevention of Cardiovascular Disease: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2019 Sep 10;74(10):1376-1414. doi: 10.1016/j.jacc.2019.03.009. Epub 2019 Mar 17. PMID 30894319
- [Background] Kong W, Wei J, Abidi P, Lin M, Inaba S, Li C, Wang Y, Wang Z, Si S, Pan H, Wang S, Wu J, Wang Y, Li Z, Liu J, Jiang JD. Berberine is a novel cholesterol-lowering drug working through a unique mechanism distinct from statins. Nat Med. 2004 Dec;10(12):1344-51. doi: 10.1038/nm1135. Epub 2004 Nov 7. PMID 15531889
- [Background] Chang W, Chen L, Hatch GM. Berberine as a therapy for type 2 diabetes and its complications: From mechanism of action to clinical studies. Biochem Cell Biol. 2015 Oct;93(5):479-86. doi: 10.1139/bcb-2014-0107. Epub 2014 Dec 1. PMID 25607236